CLINICAL TRIAL: NCT05194267
Title: Intensive Transcranial Direct Current Stimulation in the Treatment of Major Depression: Feasibility Study
Brief Title: Intensive tDCS for MDD: Feasibility Study
Acronym: tDCSintensif
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-9546
Record Dates: First submitted 2021-12-16; First posted 2022-01-18 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Open label feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active tDCS (Experimental): Will be receiving active intensive tDCS treatment
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS alters brain excitability using a weak electric field induced through two electrodes and could potentially improve symptoms of depression

SUMMARY:
This will be a prospective, open-label, single-arm study to determine the safety and feasibility of an intensive treatment of transcranial direct current stimulation (tDCS) for major depressive disorder (MDD). Participants will be age 18-65 with a diagnosis of unipolar MDD. Participants will receive an intensive treatment of tDCS over a 10-day treatment period and complete follow-up assessments at the end of treatment, 1, and 4 weeks post-treatment.

DETAILED DESCRIPTION:
This will be a prospective, open-label, single-arm study to determine the safety and feasibility of an intensive treatment of transcranial direct current stimulation (tDCS) for major depressive disorder (MDD). Secondary objective is to gather preliminary data on the clinical effects of the protocol. After assessment and inclusion into the study, participants will receive up to 50 tDCS sessions over 10 days.

Study procedures:

Daily assessments: brief questions before and after each tDCS session to evaluate potential adverse events as well as a verbal rating scale for pain.

Questionnaires : a battery of mood questionnaires will be completed to inform findings regarding clinical effects of the treatment.

Cognitive measures: a short cognitive assessment will be completed to inform findings regarding cognitive safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major unipolar depression for at least 4 weeks meeting the criteria of the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5)
* Age between 18 to 65
* Minimum score of 17 on the GRID-Hamilton Depression Rating Scale (GRID-HAMD)

Exclusion Criteria:

* Bipolar disorder,
* Psychosis
* Active substance use disorder (in the last 3 months)
* Personality disorder
* Neurocognitive disorder
* High risk of suicide
* Major comorbid medical or neurological condition
* Pregnancy

Medical contraindications to tDCS:

* Ferromagnetic material in the skull
* Defect in the bone substance of the skull
* Dermatological condition (e.g. eczema, psoriasis, urticaria, dermatitis, acne, hyperhidrosis, folliculitis, rosacea, keratosis, herpes, infectious or neoplastic phenomenon, etc.)
* Skin lesion on the skull (ex: cuts, abrasions, rash, tattoos on the skull, piercings on the head, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Miron, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS
Started | 30
Completed | 28
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Active tDCS
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Mean (Standard Deviation); unit: years] | 15.4 (2.1)
Length of current depressive episode [Mean (Standard Deviation); unit: months] | 14.4 (9.6)
Age at first depressive episode [Mean (Standard Deviation); unit: years] | 26.9 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms Measured by the Patient Health Questionnaire (PHQ-9)
Description: This outcome reflects the percentage change in depressive symptom severity as measured by the Patient Health Questionnaire-9 (PHQ-9), a 9-item self-report scale assessing depressive symptoms over the past 2 weeks. Each item is scored from 0 ("Not at all") to 3 ("Nearly every day"), with a total score ranging from 0 to 27. Higher scores indicate more severe depression. Percentage change from baseline (T0) was calculated at two follow-up timepoints:
  * T1 = 1 week after end of treatment (Day 17)
  * T2 = 1 month after end of treatment (Day 40) Percentage change was calculated using the formula: ((T_follow-up - T0) / T0) × 100. A negative value indicates improvement.
Time Frame: T0 (baseline), T1 (1 week after end of treatment) and T2 (one month after the end of the treatment)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Active tDCS
Number analyzed (Participants) | 28
percentage of change
  T1 | 21 (31.9)
  T2 | 31.5 (34.8)

ADVERSE EVENTS:
Time Frame: From Day 1 of treatment (T0) to one-month post-treatment follow-up (T2, Day 40)
Description: Same definition than from clinicaltrials.org
Arm/Group | Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 28/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS (N=28)
Tingling, itching, or burning sensation during stimulation (Skin and subcutaneous tissue disorders) | 28
Skin redness after stimulation (Skin and subcutaneous tissue disorders) | 28
Headache (Nervous system disorders) | 19
Contact dermatitis (Skin and subcutaneous tissue disorders) | 18
Fatigue (General disorders) | 16
Burning sensation (Skin and subcutaneous tissue disorders) | 7
Dizziness/light-headedness (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 3
Electric shock-like sensations (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT05194267/Prot_SAP_000.pdf